CLINICAL TRIAL: NCT02491242
Title: The Efficacy and Safety of Dolutegravir-based Dual Therapies in HIV-infected Patients With Intolerance or Toxicity to Nucleoside Analogues
Brief Title: Dolutegravir-based Dual Therapies in HIV-infected Patients With Virological Suppression
Acronym: DOLBI
Status: Completed | Type: Observational
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Responsible Party: Principal Investigator, Jose L. Casado, Physician, MD, PhD, Asociacion para el Estudio de las Enfermedades Infecciosas
Other Study IDs: Dolbi
Record Dates: First submitted 2015-06-28; First posted 2015-07-08 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: HIV Infection
Keywords: HIV; dolutegravir; intolerance; dual therapies
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Dolutegravir in a dual therapy regimen — None. Patients initiating Dolutegravir-based dual therapy because of nucleoside analogues toxicity or intolerance will be followed up during a year

SUMMARY:
The objective of this study was to evaluate the efficacy and safety, and evolution of causes leading to change, of dual therapies based in Dolutegravir in patients requiring a change of virologically effective antiretroviral therapy.

DETAILED DESCRIPTION:
Despite the high rate of virological suppression and low risk of toxicity, HIV-infected patients continue to need new antiretroviral strategies, such as dual therapies, because of different end-organ involvement (kidney, bone, cardiovascular..), intolerance or toxicity. To date, only a protease inhibitor (PI)-based regimen was able to permit the use of dual therapies (two antiretrovirals), especially in case of patients with history of virological failure to other regimens. However, the recent license of Dolutegravir, a integrase inhibitor with high genetic barrier, could help to clinicians to manage patients with intolerance or toxicity to nucleoside analogues without putting in risk virological suppression.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Receiving a virologically effective antiretroviral regimen
* Switching to a dual therapy based in dolutegravir because of intolerance or toxicity to nucleoside analogues

Exclusion Criteria:

* Pregnant women
* Receiving other investigational drugs
* Recent diagnosis of opportunistic infection (< 1 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients who had initiate a dolutegravir-based dual therapy because of intolerance or toxicity to nucleoside analogues
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Efficacy, measured as maintenance of virological suppression, after switching to a dolutegravir-based dual therapy | 12 months
  Percent of patients remaining with HIV RNA level below 50 copies/ml, according to a missing=failure criteria

SECONDARY OUTCOMES:
Safety according to DAIDS grade events 2009 of dual therapy based in dolutegravir | 12 months
  To collect adverse events (according to DAIDS grade events, 2009) and rate of discontinuation related with adverse events, of dual therapy after switching
Outcome of causes leading to switch the previous regimen | 12 months
  Evolution of causes de change: glomerular filtration rate during evolution, tubular dysfunction (proteinuria, phosphaturia, glycosuria, uricosuria),bone mineral density by DXA (dual X-ray absorptiometry), lipid disorders, adherence
Efficacy, measured as maintenance of virological suppression, of different dual therapies with dolutegravir | 12 months
  Comparison of efficacy (HIV RNA level < 50 c/ml) of the different dolutegravir-based dual therapies, according to accompanying drug (non nucleoside, especially rilpivirine), protease inhibitors (darunavir boosted with ritonavir or cobicistat), or nucleoside analogues (lamivudine).

OTHER OUTCOMES:
Rate of virological suppression in patients with previous failure to more than 2 families of antiretroviral drugs | 12 months
  Effect of extended previous failure, or mutations in the transcriptase and protease gene, in the rate of virological suppression in dolutegravir-based dual therapies

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Casado, MD, PhD, Principal Investigator — Ramon y Cajal Hospital
Locations (1):
- Ramon y Cajal Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Casado JL, Monsalvo M, Fontecha M, Vizcarra P, Rodriguez MA, Vivancos MJ, Moreno S. Dolutegravir plus rilpivirine as dual regimen in virologically suppressed HIV-1 infected patients in a clinical setting. HIV Res Clin Pract. 2019 Apr;20(2):64-72. doi: 10.1080/15284336.2019.1628460. Epub 2019 Jun 19. PMID 31303142
- [Derived] Vizcarra P, Fontecha M, Monsalvo M, Vivancos MJ, Rojo A, Casado JL. Efficacy and safety of dolutegravir plus boosted-darunavir dual therapy among highly treatment-experienced patients. Antivir Ther. 2019;24(6):467-471. doi: 10.3851/IMP3319. PMID 31172977